CLINICAL TRIAL: NCT00465387
Title: Falls, Fracture, and Osteoporosis Risk Control Evaluation (FORCE) Study: A Randomized Controlled Trial With Community Partnerships in Northern Ontario
Brief Title: FORCE (Falls, Fracture, and Osteoporosis Risk Control Evaluation) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Group Health Centre (Other)
Collaborators: Sault Area Hospital (Other); Algoma Community Care Access Centre (Other); Pharma Companies Alliance (Aventis and Proctor & Gamble) (Unknown); Merck Frosst Canada Ltd. (Industry); Eli Lilly and Company (Industry); The Green Shield Foundation (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FORCE1234
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Accidental Falls; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Falls, Fractures & Osteoporosis Risk Assessment & Management

SUMMARY:
Falls and osteoporosis-related fractures cause substantial morbidity and mortality in the elderly, and are an increasingly important public health concern. A comprehensive multidisciplinary and integrated community-based approach is needed to identify and manage the population at highest risk of these complications. Unfortunately, current gaps in continuity of care and health intervention result in a sub-optimal state of health service for these individuals. The Falls, Fracture and Osteoporosis Risk Control and Evaluation (FORCE) Study is a two-year randomized controlled trial evaluated on the effect of coordinated community-based, multidisciplinary approach for fall and fracture prevention in Sault Ste. Marie.

DETAILED DESCRIPTION:
The FORCE partners are a broad collaboration of interested consumers, stakeholders and providers, led by the Algoma Health Unit (AHU) and the Group Health Centre (GHC) - a community-based, not-for-profit, multidisciplinary health organization. Other partners include the multi-agency, consumer-orientated Algoma District Slips, Trips and Falls Committee, the Sault Area Hospital (SAH), the Algoma Community Care Access Centre (ACCAC), and Pharma Companies Alliance (Aventis and Proctor & Gamble), Merck Frosst and Lilly. The Green Shield Foundation has also provided sponsorship.The results of this study might directly benefit up to eight thousand seniors in the district by providing the impetus to integrated, evidence-based health services. Qualitative and quantitative research during this time will also be a unique opportunity to identify the modifiable barriers to the continuity and quality of care in this high-risk population. By involving the community, the project will also educate those at future risk and hopefully prevent disease and complications. Evaluation and research should provide nationally suggestions for better health service delivery.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* independent living within the city of Sault Ste. Marie, Ontario, Canada
* capable of providing informed consent

Exclusion Criteria:

* not at risk for falls
* unable to give informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Fall risk management, assessment and management of gate, strength and balance deficits, completion of medication review, including postural hypotension and psychotropic medications as well as the assessment and management of environmental risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Ciaschini, MD, FRCPC, Principal Investigator — Group Health Centre, Sault Ste. Marie, ON, Canada; Sharon E. Straus, MD MSc FRCPC, Principal Investigator — University of Toronto, ON, Canada

REFERENCES:
- [Derived] Ciaschini PM, Straus SE, Dolovich LR, Goeree RA, Leung KM, Woods CR, Zimmerman GM, Majumdar SR, Spadafora S, Fera LA, Lee HN. Community based intervention to optimize osteoporosis management: randomized controlled trial. BMC Geriatr. 2010 Aug 27;10:60. doi: 10.1186/1471-2318-10-60. PMID 20799973
- [Derived] Ciaschini PM, Straus SE, Dolovich LR, Goeree RA, Leung KM, Woods CR, Zimmerman GM, Majumdar SR, Spadafora S, Fera LA, Lee HN. Community-based randomised controlled trial evaluating falls and osteoporosis risk management strategies. Trials. 2008 Nov 4;9:62. doi: 10.1186/1745-6215-9-62. PMID 18983670
- See also: Group Health Centre website — http://www.ghc.on.ca